CLINICAL TRIAL: NCT02522117
Title: Effectiveness of Atorvastatin on IL2, IL6, TNFalpha and HLA Levels in the Recipient's Kidney Graft From a Living Donor
Brief Title: Atorvastatin in the Recipient's Kidney Graft From a Living Donor
Acronym: ATORV15
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, CLOTILDE FUENTES OROZCO, PhD, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2013-1301-100
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Renal Insufficiency
Keywords: Kidney Transplantation; Atorvastatin; Human Leukocyte Antigens; Interleukin
MeSH Terms: conditions — Renal Insufficiency | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): 24 patients received oral atorvastatin 40 mg once a day, for 4 weeks.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): 24 patients received oral placebo 40 mg once a day, for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Patients were assigned to two groups; one of them received oral atorvastatin (study group), and the other homologated placebo (control group) for 4 weeks before transplant. Then IL2, IL6, TNFalpha and HLA levels were assessed in the recipient's kidney graft by visual analog scale at prior reperfusion, and after 3 and 12 months.
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo — Patients were assigned to two groups; one of them received oral atorvastatin (study group), and the other homologated placebo (control group) for 4 weeks before transplant. Then IL2, IL6, TNFalpha and HLA levels were assessed in the recipient's kidney graft by visual analog scale at prior reperfusion, and after 3 and 12 months.
  Other Names: Homologated placebo
  Arms: Placebo

SUMMARY:
Renal insufficiency is a priority disease in the health system, which may require renal replacement therapy based on kidney transplantation, which is considered as therapy of choice. During the procedure of kidney transplantation, the body is subjected to ischemia-reperfusion damage that generates late complications related to graft function.

Recently the anti-inflammatory and immunomodulatory effects of statins have been emphasized, which could be beneficial in kidney transplantation.

DETAILED DESCRIPTION:
Objective: Evaluate the effect of atorvastatin on IL2, IL6, TNFalpha and HLA levels in the recipient's kidney graft from a living donor.

Material and methods: Controlled, double-blind trial with 12 months follow-up. Composed of 48 patients, randomized manner, realized at the Transplant Department of Western Medical Center, Mexican Institute of Social Security. Universe was patients accepted as kidney donors and their recipients. Patients included as donors were randomized into two groups (study or control) the intervention was implemented 4 weeks before kidney transplant. During surgical procedure, a biopsy from the recipient's kidney graft was obtained to measure IL-2, IL-6 TNFalpha and HLA by immunohistochemistry, 3 and 12 months after surgery. Recipients kidney function, surgical complications and kidney graft survival were registered. During surgical procedure, 3 and 12 months of following, biopsies were obtain to performed histopathological analysis based on Banff classification of renal allograft rejection grades.

The statistical analysis was performed according to the nature of variables, for continuous data using measures of central tendency and dispersion and for the qualitative data with frequencies and percentages. Inferential analysis with student's t-test, and/or Mann-Whitney's U test; chi-square distribution, and/or Fisher's exact test respectively.

ELIGIBILITY:
Donors Inclusion Criteria:

* Accepted as kidney donor
* Voluntary participation
* Informed consent accepted
* 85% fulfillment of atorvastatin treatment
* Entitlement to the Mexican Institute of Social Security

Donors Exclusion Criteria:

* Hypersensibility to Atorvastatin
* Smoking

Recipients Inclusion Criteria:

* Accepted as kidney recipient
* Entitlement to the Mexican Institute of Social Security

Recipients Exclusion Criteria:

* Patients who dropped out from study or withdrew the informed consent
* Insufficient kidney biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
HLA levels in the kidney graft biopsy | 12 months
  HLA levels were measure by immunohistochemistry, observing alteration between groups.

SECONDARY OUTCOMES:
Renal function | 12 months
  In a blood sample and in a urine 24-hour collection, serum creatinine, serum urea, creatinine clearance, urine output, and proteinuria were measure. Differences in evolution and alteration between the 2 groups were registered.
Kidney graft survival | 12 months
  In a renal biopsy using the Banff classification of renal allograft rejection grades, were assessed histologic and molecular features by microscopy and immunofluorescence. Alterations between groups were registered.
Surgery complications | 12 months
  During surgical procedure and following, any kind of complication was registered.
TNFalpha levels in the kidney graft biopsy | 12 months
  TNFalpha levels were measure by immunohistochemistry, observing alteration between groups.
IL2 and IL6 levels in the kidney graft biopsy | 12 months
  IL2 and IL6 levels were measure by immunohistochemistry, observing alteration between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde Fuentes-Orozco, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco, Mexico